CLINICAL TRIAL: NCT00559208
Title: The Comparative Effects and Expense of Augmenting Usual Children's Aid Society (CAS) Care With a Regional Differential Response and Wraparound Prevention Service for Children
Brief Title: Children's Aid Societies: Differential Response and Wraparound Prevention Trial
Status: Completed | Type: Observational
Sponsor: Hamilton Children's Aid Society (Other)
Collaborators: McMaster University (Other)
Responsible Party: Dominic Verticchio, Hamilton Children's Aid Society
Other Study IDs: 06-103; NCT00397085 (Other Grant/Funding Number: Ministry of Children & Youth Services); NCT00397085 (obsolete NCT alias)
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2009-11

CONDITIONS: Children
Keywords: Children and Youth; Families; Differential Response

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Children's Aid Societies: Comparing differential response (Wraparound) with usual care

SUMMARY:
The purpose of this study is to assess the cost-effectiveness of this Differential Wraparound model, in 5 Children's Aid Societies within Hamilton-Niagara Region, in preventing maltreatment cases from either becoming ongoing protection cases, or the children ending up in out-of-home of out-of community placements, as well as reducing the amount of time in Children's Aid Society care as compared to usual Children's Aid Society risk assessment and protection service alone.

DETAILED DESCRIPTION:
The number of children in child welfare care has increased from 10,000 in the early 1990s to over 18,000. Ontario spends over $1.1 billion a year on direct child welfare services, more than twice as much as spent in the late 1990s, with the majority of these resources spent on investigation instead of treatment. In response to this situation, Differential Response models, sometimes called alternative, multiple or integrated system responses, have been implemented in the US, Australia and Canada and are all at the beginning stages of systematic evaluation. These models will help prevent maltreatment cases from becoming ongoing protection cases, or the children ending up in out of home or community placements, and reduce the amount of time in Children's Aid Society care. This research will show the benefits and costs of a Differential Response approach to Children's Aid Society care, specifically in the Hamilton-Niagara Region

ELIGIBILITY:
Inclusion Criteria:

* Parent of children and youth, living in Hamilton and surrounding areas.
* Newly referred substantiated cases going on to protective services.
* English & non-English speaking.

Exclusion Criteria:

* Safety threat
* Non-substantiated cases not going to protective services.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clients of CAS going on to protective custody cases
Sampling Method: Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2006-10; Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To measure the characteristics of families and their children and comparisons between usual care versus differential response | Follow-up at 1 year and 2 years

SECONDARY OUTCOMES:
Follow up measures at 1 year and 2 year follow ups including measuring whether differential response is happening | 6 months after facilitator is assigned

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Verticchio, Principal Investigator — Children's Aid Society
Locations (1):
- Children's Aid Society, Hamilton, Ontario, Canada